CLINICAL TRIAL: NCT01693809
Title: The Effects of Caffeine on Vestibular Evoked Myogenic Potentials in Healthy
Brief Title: The Effects of Caffeine on Vestibular Evoked Myogenic Potentials in Healthy Subjects
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital do Servidor Publico Estadual (Other)
Responsible Party: Principal Investigator, Ana Maria Almeida de Sousa, MD, Hospital do Servidor Publico Estadual
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: 0127/11
Record Dates: First submitted 2012-09-20; First posted 2012-09-26 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Healthy Subjects
Keywords: Caffeine; Vestibular Evoked Myogenic Potentials; dizziness; vertigo; tinnitus
MeSH Terms: conditions — Dizziness; Vertigo; Tinnitus | interventions — Caffeine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Caffeine (Experimental): Caffeine 420mg, one time
  Interventions: Drug: Caffeine

INTERVENTIONS:
Drug: Caffeine

SUMMARY:
The principal aim of this study is to evaluate the presence of changes in cervical vestibular evoked myogenic potentials (VEMPc) after acute intake of caffeine in healthy subjects.

Secondarily, it wants to standardize normal values exam VEMPc in otorhinolaryngology service of the hospital.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* hearing impairment
* caffeine abuse 24 hours before the test
* medication remains
* hypertension, dyslipidemia, diabetes mellitus or sleep disorders.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-10 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Alteration of p13 and n23 latency and p13-n23 amplitude before and after caffeine intake. | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Akira Suzuki, PhD, Study Chair — Hospital do Servidor Publico Estadual; Ana Maria Almeida Sousa, MD, Principal Investigator — Hospital do Servidor Publico Estadual
Locations (1):
- Hospital do Servidor Publico Estadual, São Paulo, São Paulo, Brazil